CLINICAL TRIAL: NCT04130763
Title: Investigator-initiated Trial of Fecal Microbiota Transplant (FMT) Capsule for Improving the Efficacy of Anti-PD-1 in Patients with PD-(L)1 Resistant Digestive System Cancers
Brief Title: Fecal Microbiota Transplant (FMT) Capsule for Improving the Efficacy of Anti- PD-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XBI-302CT1001
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Gastrointestinal System Cancer
Keywords: Immuno-checkpoint inhibitor therapy; GI cancer; FMT
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMT Capsule in Combination with Anti-PD-1 Therapy (Experimental): FMT Capsule in Combination with Anti-PD-1 Therapy
  Interventions: Biological: FMT capsule

INTERVENTIONS:
Biological: FMT capsule — FMT capsules administration starts in the first week of enrollment. Capsules are taken for three consecutive days in the first week. From week 2, anti-PD-1 therapy will be administrated in combination with the maintenance dose of FMT treatment once every two weeks for up to 6 times.

SUMMARY:
To determine whether the fecal microbiota transplant (FMT) capsule can help reverse the resistance of anti-PD-(L)1 treatment in Gastrointestinal (GI) cancer patients.

DETAILED DESCRIPTION:
This study is designed to improve the response rate of anti-PD-(L)1 among patients with anti-PD-(L)1 resistant/refractory digestive (including gullet, stomach and intestine) system cancers through the intervention on their gut microbiota. Healthy people who have the gut microbiota profile similar to the responders of anti-PD-(L)1 therapy will be identified. The gut microbiota of these healthy people will be extracted to product FMT capsule. Gastrointestinal (GI) cancer patients who failed anti-PD-(L)1 treatment will be administrated with anti-PD-1 immunotherapy combined with FMT. The enrolled subjects will firstly receive 1-week of FMT therapy. Subsequently, each anti-PD-1 treatment will be combined with the maintenance dose of FMT capsules to ensure the efficiency of gut microbiota colonization. Each subject will receive anti-PD-1 therapy for 6 cycles. After the completion of both 3 and 6 cycles of therapy, safety and efficacy assessments will be conducted. The subjects who complete 3 cycles of treatment but are clinically evaluated as disease progression will not continue to the following 3 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient had a histologically or cytologically confirmed diagnosis of unresectable or metastatic solid tumors originating from the GI tract.
2. Patient was able and willing to provide pathological tissue embedded in wax blocks or paraffin sections.
3. Patient had received any number of radiation therapy, chemotherapy, vaccine therapy or other oncological therapy are permitted.
4. Patient was receiving or has received at least 2-dose injections of systemic PD-(L)1 immunotherapy, and imaging results confirmed progressive disease (PD). According to iRECIST, PD is defined as an increase in the length of the lesion > 20% or occurrence of new lesion or non-target lesion progression. Anti-PD-(L)1 drugs can contain pembrolizumab, nivolumab or any other anti-PD-(L)1 drugs that have passed phase 2 clinical development. Patients are eligible when the previous failed anti-PD-(L)1 treatment was initiated within one year of the first dose of this trial.
5. Patient was willing and able to swallow at least 20 FMT capsules.
6. Patient was willing and able to sign the informed consent form.
7. Patient consented to receive follow-up medical imaging to determine disease progression and provide stool samples before and after taking capsules at each follow-up visit.
8. Patient was at least 18 years old, male or female.
9. Patient had an ECOG performance of 0 or 1.
10. For women with childbearing potential, the results of blood pregnancy test within 7 days prior to enrollment or the results of urine pregnancy test within 72 hours prior to enrollment had to be negative.
11. Patient must have had basic body function. Blood test results needed to reach the following indexes: Absolute neutrophil count (ANC)≥1500/mcL, platelets≥100,000/mcL, hemoglobin≥9 g/dL or 5.6 mmol/L, no transfusion or EPO dependency (within 7 days of assessment), serum creatinine≤1.5×upper limit of normal (ULN) or creatinine clearance≥60 mL/min, serum total bilirubin≤1.5×ULN or direct bilirubin≤ULN, AST (SGOT) and ALT (SGPT)≤2.5×ULN for patients with serum total bilirubin >1.5 ULN or ≤5×ULN for patients with liver metastases, albumin≥2.5 mg/dL, coagulation indexes INR or PT ≤1.5×ULN. Unless patient was receiving anticoagulant therapy, coagulation indexes were within normal range of therapy.
12. Expected survival duration ≥3 months.

Exclusion Criteria:

1. Patient with irritable bowel syndrome, toxic megacolon, and severe dietary allergies (including severe allergic to shellfish, nuts, seafood).
2. Patient had responded to anti-PD-(L)1 therapy or had a stable disease status (per iRECIST at CR, PR, or SD).
3. Patient had participated in any other clinical trial within 4 weeks before the first dose of FMT capsule treatment.
4. Patient had highly severe symptoms including rapidly declining ECOG performance; rapidly worsening symptoms; lesion transferring to critical sites and requiring urgent medical intervention.
5. Patient had a known history of malignant blood diseases, primary brain tumor or sarcoma, or other primary solid tumors except gastrointestinal tumors.
6. Patient had progressing CNS metastases or leptomeningeal metastases. Patients with stable brain metastases had to be re-screened by brain MRI or CT scan within two weeks before enrollment to ensure no disease progression, and simultaneously take ≤10mg steroid daily one week prior to treatment. Patients with no history of CNS metastases and no signs of CNS metastases did not need another medical imaging examination for brain diseases.
7. Patient had a severe hypersensitivity or reaction to anti-PD-(L)1 immunotherapy.
8. Patient had an autoimmune disease or a history of autoimmune disease or required treatment with systemic steroid (prednisone >10 mg daily or equivalent dose of similar drugs) or immunosuppressive agents. The following cases were exceptions: local, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with extremely low systemic absorption; hormone replacement therapy; short-term (≤7 days) treatment of corticosteroids for preventative use (e.g., allergy to contrast agents).
9. Patient had pneumonitis or had a history of (non-infectious) pneumonitis requiring steroid therapy.
10. Patient had severe cardiovascular disease (e.g., drug-uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, severe obstructive or restrictive pulmonary diseases, or systemic infections.
11. Patient had active human immunodeficiency virus (HIV) infection (performance as HIV 1/2 antibodies and/or positive).
12. Patient had active Hepatitis B (HBV) or Hepatitis C (HCV) infection.
13. Patient had known active tuberculosis.
14. Patient had received a live vaccine or live attenuated vaccine within 4 weeks prior to enrollment.
15. Patient had reported adverse events (per CTCAE 5.0, ≥grade 2) due to drug treatment within 4 weeks and not recovered from it. Patients who had undergone major surgery had to have completely recovered from toxicity and complications of previous interventions prior to participating in the study.
16. Patient had received anti-tumor therapy except experimental drugs (e.g., chemotherapy, targeted small molecule therapy or radiotherapy) within 2 weeks prior to screening or planned to receive anti-tumor therapy except experimental drugs (e.g., chemotherapy, targeted small molecule therapy or radiotherapy) during the study period. Radiotherapy used for pain control was an exception.
17. Patient had a known history of psychiatric disorders or drug abuse.
18. Patient was pregnant or breastfeeding, or subjects (including male subject and his female spouse) could not take effective contraceptive measures at the time of signing the informed consent until 120 days after the final anti-PD-1 therapy combined with FMT treatment.
19. Patient could not stop antibiotics treatment 24 hours before administration due to infection, etc.
20. Other cases that investigators qualified as relevant for patients who could not participate in the study, e.g., any medical history, treatment history, or history of abnormal test data that possibly confuses the study results, or interferes with patients' participation in the whole study, or damages patient interests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 14 weeks
  Number of subjects with objective responses (Complete Response (CR) + Partial Response (PR)) divided by total number of subjects, per iRECIST.
The number of adverse events | 1 week
  The number of adverse events that is related to FMT prior to the first anti-PD-1 immunotherapy treatment.
Rate of abnormal vital signs and laboratory test results | 1 week
  Rate of abnormal vital signs and laboratory test results that are determined to be clinically significant prior to the first anti-PD-1 immunotherapy treatment.

SECONDARY OUTCOMES:
Change in T-cells Composition | 14 weeks
  Compare the changes in CD8+PD-1+T cells, Ki67+CD8+ T cells before and after treatment between response subjects and non-response subjects (evaluated by iRECIST).
Function of T-cells | 14 weeks
  Compare the changes in cells expressing IFN-γ before and after treatment between response subjects and non-response subjects (per iRECIST).
Association of anti-PD-1 response with gut microbiota | 14 weeks
  Compare the changes in bacterial abundance and bacterial diversity before and after treatment between response subjects and non-response subjects (per iRECIST).
Rate of abnormal vital signs, physical examination results, 12-lead electrocardiogram and laboratory test results | 14 weeks
  Rate of abnormal vital signs, physical examination results, 12-lead electrocardiogram and laboratory test results that are determined to be clinically significant from the beginning of the first anti-PD-1 immunotherapy treatment to the end of study.
Change in subsets of specific and non-specific immune system | 14 weeks
  Compare the changes in T-cell receptor diversity (quantified by immune repertoire sequencing analyses), CD8+CCR7+CD45RA+T cells, CD4+CCR7+CD45RA+ T cells ,CD4 + Foxp3 + T cells,CD56+NK cells and CD68+ cells before and after treatment between response subjects and non-response subjects (evaluated by iRECIST).
The number of adverse events | 14 weeks
  The number of adverse events from the beginning of the first anti-PD-1 immunotherapy treatment to the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No